CLINICAL TRIAL: NCT02785965
Title: Acupuncture in the Regulation of Dai Meridian for Polycystic Ovarian Syndrome Patients With Abdominal Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Dongfang Hospital Beijing University of Chinese Medicine (Other)
Collaborators: Beijing University of Chinese Medicine (Other); Beijing Municipal Science & Technology Commission (Other)
Responsible Party: Principal Investigator, Hui Hu, Director,clinical research, Dongfang Hospital Beijing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Z161100000516057
Record Dates: First submitted 2016-05-23; First posted 2016-05-30 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Polycystic Ovarian Syndrome; Obesity, Abdominal
Keywords: electroacupuncture; lifestyle modification; diet; exercise; Dai Meridian
MeSH Terms: conditions — Polycystic Ovary Syndrome; Obesity, Abdominal; Motor Activity | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- acupuncture & lifestyle modification (Experimental): Electro-acupuncture is given three times a week with diet restriction to 1400 calories a day and moderate aerobic exercise 3h a week for 12 weeks.
  Interventions: Device: electroacupuncture; Behavioral: lifestyle modification
- lifestyle modification (Active Comparator): diet restriction to 1400 calories a day and moderate aerobic exercise 3h a week for 12 weeks
  Interventions: Behavioral: lifestyle modification

INTERVENTIONS:
Device: electroacupuncture — Disposable, single-use, sterilized stainless-steel needles (Yunlong, Beijing, China; length 40/100 mm, diameter 0.30 mm) are inserted into waist, bilaterally. All of the six points are located in the Dai Meridian route corresponding to the ovaries. Four needles, 0.25mm in diameter and 25mm in length, are also placed in distal acupuncture points which are located in the feet and lower arms to enhance local points' effects. Acupuncture needles of 0.3mm in diameter and 100mm in length are inserted into GB26(Daimai) with a depth of 25-65mm by an angle of 15°, following the path of Dai Meridian (towards medial and downside). The other needles are inserted vertically into the acupoints with a depth of 10-30mm, depending on the thickness of muscles. Electro-acupuncture is applied to both sides of GB26 and ST25(Tianshu): cathode is connected to GB26; anode to ST25. Needles are stimulated electrically with low frequency (2 Hz) for 20 min.
  Arms: acupuncture & lifestyle modification
Behavioral: lifestyle modification — The diet restricts patients to 1400 calories a day for 12 weeks.The exercise included 12 weeks of aerobic exercise in moderate level (60 to 70% of maximum heart rate), for 3 sessions a week, each session for 60 min. The exercises included: Warning up: 10 min, main phase (aerobic exercise): 40 min and cooling down: 10 min. Polar Pulse measuring device from China was used to control the intensity of the exercises.

SUMMARY:
The purpose of this study is to determine whether the use of electroacupuncture to dredge and regulate Dai Meridian combined with lifestyle modification are more effective than lifestyle modification only in the treatment of anovulation and hyperandrogenism due to polycystic ovary syndrome (PCOS) with abdominal obesity.Two thirds of participants will receive electroacupuncture and lifestyle modification in combination, while the other one third will receive lifestyle modification only.

DETAILED DESCRIPTION:
Obesity, especially abdominal obesity, is one of most common clinical features of polycystic ovary syndrome, a widely and seriously influenced complex disorder related to reproduction and metabolism. Excessive accumulation of adipose tissue in the abdominal organs often leads to insulin resistance, which will increase the harm of hyperandrogenism and exacerbate ovulation disorders and metabolic abnormalities.

Weight loss, likely beneficial for both reproductive and metabolic dysfunction in this setting , has been generally recommended as a first-line therapy for obese women with PCOS and can be accomplished via lifestyle modification and electroacupuncture. What's more, stimulating acupoints of Dai Meridian can regulate menstrual cycles and treat infertility according to the theory of traditional Chinese medicine. However, how much benefits patients will additionally get from the Combined therapy is not clear now.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Polycystic Ovarian Syndrome.
* Clinical diagnosis of abdominal obesity.
* Agree to participate in clinical trials.

Exclusion Criteria:

* Endocrine or neoplastic causes of amenorrhoea, anovulation and hyperandrogenemia, including central nervous system abnormalities, premature ovarian failure, thyroid disease, Cushing's syndrome,androgen secreting tumors, congenital adrenal hyperplasia, and hyperprolactinaemia.
* Patients suffering from other serious diseases(cardiocerebrovascular diseases, damage to the function of liver and kidney, and mental illness).
* Patients taking hormonal and metabolic drugs within 12 weeks of study entry affecting the judgment of results.
* Pregnant or breast feeding.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-01 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
rate of recovered ovulation | 12 weeks
  the proportion of patients who have ovulation after treatment

SECONDARY OUTCOMES:
evidence of clinically definite hyperandrogenism confirmed by mF-G score | 12 weeks
evidence of clinically definite hyperandrogenism confirmed by the Global Acne Grading System | 12 weeks
frequency of menstruation | 12 weeks
quantity of menstruation | 12 weeks
  pictorial blood loss assessment chart
Serum total testosterone (T) | 12 weeks
FSH | 12 weeks
  follicle stimulating hormone (FSH)
LH | 12 weeks
  luteinizing hormone (LH)
ovarian volume measured by ultrasound | 12 weeks
follicle number pre ovary measured by ultrasound | 12 weeks
ovarian stromal blood flow measured by ultrasound | 12 weeks
body weight in kilograms | 4, 8 and 12 weeks
waist circumference in centimeter | 4, 8 and 12 weeks
BMI in kg/m^2 | 4, 8 and 12 weeks
waist-to-height ratio | 4, 8 and 12 weeks
  waist-to-height ratio=waist circumference in centimeter/height in centimeter
Fasting serum PAI-1 level | 12 weeks
International physical activity scale (IPAQ) short version | 4, 8 and 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Hui HU, Doctor, Principal Investigator — Dongfang Hospital Beijing University of Chinese Medicine
Locations (2):
- China (2):
  - Department of Acupuncture and Moxibustion, Dongfang Hospital, Beijing University of Chinese Medicine, Beijing, Beijing Municipality
  - Dongfang Hospital Affiliated to Beijing University of Chinese, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abazar E, Taghian F, Mardanian F, Forozandeh D. Effects of aerobic exercise on plasma lipoproteins in overweight and obese women with polycystic ovary syndrome. Adv Biomed Res. 2015 Mar 25;4:68. doi: 10.4103/2277-9175.153892. eCollection 2015. PMID 25878993
- [Background] Case problem: dietary recommendations to combat obesity, insulin resistance, and other concerns related to polycystic ovary syndrome. J Am Diet Assoc. 2000 Aug;100(8):955-7; discussion 957-60. doi: 10.1016/S0002-8223(00)00275-3. No abstract available. PMID 10955058